CLINICAL TRIAL: NCT04323670
Title: BIO|MASTER.Selectra 3D Study
Brief Title: Master Study Investigating the Guiding Catheter Selectra 3D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BA110
Record Dates: First submitted 2020-03-17; First posted 2020-03-26 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2022-05

CONDITIONS: Pacemaker DDD

STUDY DESIGN:
Intervention Model Description: Guiding catheter Selectra 3D
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Selectra 3D (Other): Guiding catheter to position the brady lead into a untypical heart position
  Interventions: Device: "Selectra 3D" guiding catheter

INTERVENTIONS:
Device: "Selectra 3D" guiding catheter — His lead measurements

SUMMARY:
Study investigating the guiding catheter Selectra 3D

DETAILED DESCRIPTION:
The guiding catheter 'Selectra 3D' is a catheter that is intended to support the implantation of a pacemaker lead in untypical positions in the heart like in the His- bundle area.

This study is designed as post market clinical follow-up (PMCF) study to identify and evaluate residual risks associated with the use of the guiding catheter Selectra 3D that remained unrevealed even after risk analysis, risk mitigation and successful conformity assessment. Moreover, the study aims at providing additional PMCF data, as required by regulatory authorities. Furthermore, the performance and efficacy of the Selectra 3D shall be assessed. The results will be used for updating the clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Standard indication for de novo pacemaker or cardiac resynchronization implantation
* The patient is intended for guiding catheter based implantation of a pacemaker system
* Patient is able to understand the nature of the study and has provided written informed consent
* Patient is willing and able to perform all follow up visits at the study site
* Patient is willing and able to use the CardioMessenger and accepts the BIOTRONIK Home Monitoring® concept

Exclusion Criteria:

* AV block with no escape rhythm or broad QRS escape rhythm
* Standard contraindications for use of the investigational devices:
* Existing or possible occlusion of the coronary vessels or unsuitable anatomy of the coronary veins
* Active systemic infection
* Mechanical tricuspid valve prosthesis or severe tricuspid valve diseases
* Intolerance against dexamethasone acetate
* Planned cardiac surgical procedures or interventional measures in addition to the study procedure within the next 6 months
* Expected to receive heart transplantation or ventricular assist device within 1 year
* Patient is pregnant or breast feeding
* Less than 18 years old
* Participating in another interventional clinical investigation
* Life-expectancy is less than 1 year

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Selectra 3D-related SADE-free rate | 7 days after implantation
  Selectra 3D-related Serious adverse device effect rate

SECONDARY OUTCOMES:
Successful implantation rate | At the day of implantation
  Assessment, if the pacemaker lead is positioned successfully in the intended target position
Appropriateness of sensing and pacing of Solia S | 12 months
  Investigator assessment for leads in His position
SADE-free rate of Solia S | 6 months
  Safety of Solia S in His position
SADE-free rate of Solia S | 12 months
  Safety of Solia S in His position

CONTACTS AND LOCATIONS:
Overall Officials: Uwais Mohamed, PhD, Principal Investigator — The Northern Hospital, Epping, Australia
Locations (1):
- CHRU de Tours, Tours, France

IPD SHARING:
Plan to Share IPD: No